CLINICAL TRIAL: NCT05228847
Title: Effect of Human Milk-derived Fortifiers on Weight Gain in Preterm Infants <1250 g: A Randomized Controlled Trial
Brief Title: Human Milk-derived Fortification in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Belal Alshaikh, Clinical Associate Professor, Department of Pediatrics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB22-039
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Postnatal Growth Restriction; Necrotizing Enterocolitis
Keywords: Human milk
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human milk-derived HMF (Active Comparator): Fortification with human milk-derived product
  Interventions: Dietary Supplement: Human milk-derived HMF
- Bovine milk-derived HMF (Other): Current standard practice: Fortification with bovine milk-derived product
  Interventions: Dietary Supplement: bovine milk-derived HMF

INTERVENTIONS:
Dietary Supplement: Human milk-derived HMF — Fortification with human milk-derived product
  Arms: Human milk-derived HMF
Dietary Supplement: bovine milk-derived HMF — bovine milk-derived HMF
  Arms: Bovine milk-derived HMF

SUMMARY:
Human Milk alone is unable to meet the high nutritional requirements of preterm infants. The American Academy of Pediatrics recommends fortification of human milk as a standard practice in all very low birth weight (VLBW) infants. Multi-nutrient human milk fortifiers (HMFs) are designed to meet the macro and micro-nutrient needs of VLBW infants. HMFs differ by the origin of milk and by nutrient composition. Traditionally, bovine milk has been the main source of multi-nutrient HMFs.

DETAILED DESCRIPTION:
Recent advances in lacto-engineering techniques allowed the manufacturing of multi-nutrient HMF from human milk as an alternative to bovine milk. Since exposure to infant bovine-based formula feeds is frequently shown to increase neonatal morbidities, human milk-derived HMFs (H-HMFs) have been frequently proposed to minimize exposure to bovine products prior to 34 weeks gestation with an intent to decrease the risks of necrotizing enterocolitis and feeding intolerance. The use of multi-nutrient H-HMFs is a promising intervention however currently available H-HMFs are expensive.

The main objective of this randomized controlled trial is to compare the weight gain achieved by preterm infants born <1250 g and fed human milk fortified with H-HMFs (made from mother's own milk (MOM) when MOM supply exceeds the daily need of her preterm infant or from donor human milk (DHM) compared with counterparts fed human milk fortified with the currently used bovine-derived fortifier (B-HMF).

ELIGIBILITY:
Inclusion Criteria:

* Birthweight between 400 g-1250 g
* Less than or 32 weeks gestational age at birth
* Subject has been classified as appropriate for gestational age
* Enteral feeding of human milk is initiated by 72 hours
* Subject is expected to be on human milk for at least 3 weeks.

Exclusion Criteria:

* Congenital abnormalities or underlying disease that may affect growth
* Maternal cocaine, alcohol, or opioid abuse during pregnancy
* Mother or infant is currently receiving treatment for HIV infection
* Infant with major surgery

Ages: 3 Days to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Average weight gain | up to 3 weeks
  Average weight gain measured as g/kg per day

SECONDARY OUTCOMES:
Head circumference | Weekly for 8 weeks
  Measurement of head circumference in centimeters
Length | Weekly for 8 weeks
  Measurement of length in centimeters
Feed intolerance | 3 weeks
  Incidence of interruption in enteral feeding due to feed intolerance (vomiting or abdominal distension), unrelated to a clinical procedure, that lasted for ≥12 hours or a >50% reduction in volume over the same time frame.
Electrolytes abnormalities | 3 weeks
  Incidence of any abnormality in one of the following electrolytes: sodium, potassium, calcium and phosphorus
Need for additional signal nutrient supplementation | 3 weeks
  Number of additions of single nutrient supplementation (include protein, fat and carbohydrate) in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada